CLINICAL TRIAL: NCT06635005
Title: A Low-Insulinemic Dietary Intervention to Reduce Breast Cancer Risk in High-Risk Women
Acronym: LIN-BRiCK
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Collaborators: American Cancer Society, Inc. (Other)
Responsible Party: Principal Investigator, Fred Tabung, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: OSU-23417; NCI-2024-08360 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2024-10-08; First posted 2024-10-10 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-10

CONDITIONS: Feasibility Pilot Study; Compliance
Keywords: Insulinemic dietary pattern, high-risk, breast cancer, cardiometabolic health
MeSH Terms: conditions — Patient Compliance; Breast Neoplasms | interventions — Specimen Handling; Diet Therapy; Motivational Interviewing; Nutrition Assessment

STUDY DESIGN:
Masking Description: This is a single arm study with a dietary pattern as intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Prevention (Low-EDIH dietary pattern intervention) (Experimental): Participants receive the low-EDIH dietary pattern intervention consisting of 6 group nutrition education sessions focusing on foods to prioritize within each food group, food combinations, food preparation, discussion, simple cooking demonstrations, food tastings, smart shopping advising, and a question/answer period over 2 hours each at weeks 0, 1, 2, 3, 5, and 6. Participants also attend 3 in-person or virtual individual nutrition counseling and motivational interviewing sessions over 30 minutes each at weeks 3 and 5, between weeks 7 and 9, and between weeks 9 and 11. Participants also wear an activity tracker and undergo blood sample collection on study.
  Interventions: Procedure: Biospecimen Collection; Other: Dietary Intervention; Other: Medical Device Usage and Evaluation; Behavioral: Motivational Interviewing; Other: Nutritional Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Other: Dietary Intervention — Receive the Low-EDIH dietary pattern intervention
  Other Names: Dietary Modification; intervention, dietary; Nutrition Intervention; Nutrition Interventions; Nutritional Interventions
Other: Medical Device Usage and Evaluation — Wear an activity tracker
Behavioral: Motivational Interviewing — Undergo motivational interviews
  Other Names: MI; Motivational Interviewing Intervention
Other: Nutritional Assessment — Participate in nutrition counseling
  Other Names: Dietary Assessment; dietary counseling; nutritional counseling
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This clinical trial tests whether a new dietary pattern that consists of foods that lower the blood insulin response can reduce breast cancer risk in high-risk women. In a large group of patients, this new dietary pattern was associated with reduced risk of multiple cancers and reduced risk of long-term weight gain. Parts of this new dietary pattern are quite different from typical dietary recommendations, and much education is needed. Overall, compared to the typical American diet, this new dietary pattern is moderately low in total fat and saturated fat, low in protein from animal foods but high in protein from plant sources, high in fruits and vegetables, high in whole grains, and high in dietary fiber. We will determine if a low-insulinemic dietary pattern intervention is feasible and effective in reducing breast cancer risk in high-risk women.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Evaluate the feasibility of translating the low-Empirical Dietary Index for Hyperinsulinemia (EDIH) dietary pattern intervention from epidemiologic cohorts to the clinic in a single arm phase I trial among postmenopausal women at high risk for cancer and evaluate safety.

SECONDARY OBJECTIVES:

I. Determine the change in patient reported outcomes (PRO) under the Low-EDIH dietary pattern at 12 weeks from baseline.

II. Evaluate the change in cardiometabolic biomarker profiles at 12 weeks from baseline (a) glycemic control and insulin response parameters measured using fasting glucose, insulin, hemoglobin A1C, C-peptide, HOMA-IR, HOMA-B and IGFBP-1, IGFBP-2, (b) lipid profiles (total cholesterol, triglycerides [TG], low density lipoprotein [LDL], higher high density lipoprotein [HDL]).

III. Assess change in circulating biomarkers associated with risk of breast cancer and low-grade chronic inflammatory state including C-reactive protein (CRP), TNFalpha-R2, IL-6 and leptin/adiponectin ratio at 12 weeks from baseline.

EXPLORATORY OBJECTIVES:

I. Collect stool samples and process for subsequent assessment of changes in the fecal microbiome structure and function related to the low-EDIH dietary pattern intervention.

II. Collect 24-hour urine samples and process for subsequent assessment of changes in targeted and non-targeted metabolomics and lipidomics alterations related to the low-EDIH dietary pattern intervention.

OUTLINE:

Participants receive the low-EDIH dietary pattern intervention consisting of 6 group nutrition education sessions focusing on foods to prioritize within each food group, food combinations, food preparation, discussion, simple cooking demonstrations, food tastings, smart shopping advising, and a question/answer period over 2 hours each at weeks 0, 1, 2, 3, 5, and 6. Participants also attend 3 in-person or virtual individual nutrition counseling and motivational interviewing sessions over 30 minutes each at weeks 3 and 5, between weeks 7 and 9, and between weeks 9 and 11. Participants also wear an activity tracker and undergo blood sample collection on the study.

After completion of study intervention, participants are followed up in week 12.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 45 years OR post-menopausal AND cis-gender women at study registration.
* Overweight or World Health Organization (WHO) class 1 obese as defined by a body mass index (BMI) of 25 to 35 kg/m^2.
* High risk for breast cancer at the discretion of the physician, using standard definitions such as a Gail 5-year risk of ≥ 2% or Tyrer Cuzick version (v) 8.0 10-year risk of ≥ 5%.
* Concurrent or prior use of endocrine therapy is allowed. Any dose or schedule change is not permitted for the duration of the study.
* Currently established care or previously seen at the Ohio State University Comprehensive Cancer Center (OSUCCC) Stefanie Spielman Comprehensive Breast Center (SSCBC) high risk breast clinic.

Exclusion Criteria:

* Prior diagnosis of breast cancer within past 5 years.
* Metastatic breast cancer (at study start or during study period).
* BMI > 35 kg/m^2 or < 25 kg/m^2.
* Pre-menopausal women or < 45 years of age.
* Assigned male at birth.
* Uncontrolled intercurrent illness including lung disease, heart disease, metabolic disease; exacerbations for disease in past 8 weeks; unstable on medications for chronic conditions in past 6 weeks. This could affect compliance and engagement with study intervention. Change in anti-hyperglycemic or lipid lowering medications is best avoided for the duration of the study unless deemed necessary by treating provider or required for acute exacerbation of existing illness.
* Type 1 diabetes mellitus (DM) or insulin dependent, or evidence of brittle diabetes.
* Presence of food allergies or intolerances to wheat, nuts, seeds, fish, or dairy foods.
* Currently on special diet for known metabolic or gastrointestinal disease, or planning to start a specific dietary regimen such as vegetarian, vegan, ketogenic, low-fat diets, etc.
* Uncontrolled psychiatric illness/social situations that would limit compliance with study requirements.
* Unwilling or unable to follow protocol requirements.
* Pregnant, trying to get pregnant, or nursing.
* Any condition which in the investigator's opinion deems the subject an unsuitable candidate to participate in this study.
* Non-English speaking, as the teaching materials and educational sessions have not yet been translated into additional languages.
* Prisoners or other institutionalized patients.

Min Age: 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Cis-gender is an inclusion criterion as hormone use may alter breast cancer risk
Enrollment: 30 (Estimated)
Dates: Start 2024-10-03 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Successful translation of the low-Empirical Dietary Index for Hyperinsulinemia dietary pattern | Up to 12 weeks
  High compliance will be defined as > 80% of participants achieving and maintaining scores ≥ median 0.06. Will be measured by the low-Empirical Dietary Index for Hyperinsulinemia scores. Descriptive statistics (i.e., means, standard deviations for continuous variables, and frequencies and percentages for discrete data) will be used to summarize demographics and clinical characteristics of study participants. Will be tested using multivariable-adjusted general linear mixed regression to accommodate within-person variance across post-baseline timepoints via a per-subject random effect. Will evaluate model assumptions via regression diagnostics and adjust model structure and outcome transformations as necessary to ensure proper model fit. Will be adjusted for age, baseline total caloric intake, body weight, and baseline value.

SECONDARY OUTCOMES:
Plasma biomarkers of cardiometabolic health | From baseline to 12 weeks
  Plasma biomarkers of cardiometabolic health include C-peptide, and IGFBP-1, IGFBP-2. Descriptive statistics (i.e., means, standard deviations for continuous variables, and frequencies and percentages for discrete data) will be used to summarize demographics and clinical characteristics of study participants. Will be tested using multivariable-adjusted general linear mixed regression to accommodate within-person variance across post-baseline timepoints via a per-subject random effect. Will evaluate model assumptions via regression diagnostics and adjust model structure and outcome transformations as necessary to ensure proper model fit. Will be adjusted for age, baseline total caloric intake, body weight, and baseline value.
Urine biomarkers of cardiometabolic health | From baseline to 12 weeks
  Descriptive statistics (i.e., means, standard deviations for continuous variables, and frequencies and percentages for discrete data) will be used to summarize demographics and clinical characteristics of study participants. Will be tested using multivariable-adjusted general linear mixed regression to accommodate within-person variance across post-baseline timepoints via a per-subject random effect. Will evaluate model assumptions via regression diagnostics and adjust model structure and outcome transformations as necessary to ensure proper model fit. Will be adjusted for age, baseline total caloric intake, body weight, and baseline value.
Patient reported outcomes (PROs) | Up to 12 weeks
  PROs will be assessed using Patient-Reported Outcomes Measurement Information System scales 29 Profile version 2.1 (domains: physical function, social roles, fatigue, depression, anxiety, pain, and sleep disturbance) and the Global Health Short Form. Descriptive statistics (i.e., means, standard deviations for continuous variables, and frequencies and percentages for discrete data) will be used to summarize demographics and clinical characteristics of study participants. Will be tested using multivariable-adjusted general linear mixed regression to accommodate within-person variance across post-baseline timepoints via a per-subject random effect. Will evaluate model assumptions via regression diagnostics and adjust model structure and outcome transformations as necessary to ensure proper model fit. Will be adjusted for age, baseline total caloric intake, body weight, and baseline value.

CONTACTS AND LOCATIONS:
Overall Officials: Fred K Tabung, PhD, MSPH, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Romanos-Nanclares A, Tabung FK, Willett WC, Rosner B, Holmes MD, Chen WY, Tamimi RM, Eliassen AH. Insulinemic potential of diet and risk of total and subtypes of breast cancer among US females. Am J Clin Nutr. 2022 Dec 19;116(6):1530-1539. doi: 10.1093/ajcn/nqac284. PMID 36178066
- [Background] Lee DH, Giovannucci EL, Tabung FK. Insulin-related dietary indices predict 24-h urinary C-peptide in adult men. Br J Nutr. 2020 Jun 19:1-8. doi: 10.1017/S0007114520002184. Online ahead of print. PMID 32618519
- [Background] Tabung FK, Wang W, Fung TT, Hu FB, Smith-Warner SA, Chavarro JE, Fuchs CS, Willett WC, Giovannucci EL. Development and validation of empirical indices to assess the insulinaemic potential of diet and lifestyle. Br J Nutr. 2016 Nov 28;116(10):1787-1798. doi: 10.1017/S0007114516003755. Epub 2016 Nov 8. PMID 27821188
- See also: The Jamesline — http://cancer.osu.edu